CLINICAL TRIAL: NCT01465412
Title: An Open-label, Single Dose, Oral Administration, Sequential Two Parts Study to Compare the Pharmacokinetics of SCH 420814 / MK-3814 in Subjects With Mild and Moderate Chronic Hepatic Impairment With Their Respectively Matching Healthy Volunteers
Brief Title: A Study to Assess Pharmacokinetics of Preladenant in Participants With Chronic Hepatic Impairment (P06513)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06513; MK-3814-034 (Other: Merck & Co.)
Record Dates: First submitted 2011-10-28; First posted 2011-11-04 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-08

CONDITIONS: Chronic Hepatic Impairment
Keywords: Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild Hepatic Impaired (HI) Part 1 (Experimental): Participants with mild chronic liver disease enrolled in Part 1 received one 5-mg preladenant tablet, orally, on Day 1.
  Interventions: Drug: Preladenant
- Healthy to Match Mild HI Part 1 (Active Comparator): Healthy volunteers with normal hepatic function matched to participants with mild chronic liver disease by race, age, BMI, and gender, enrolled in Part 1 received one 5-mg preladenant tablet, orally, on Day 1.
  Interventions: Drug: Preladenant
- Moderate HI Part 2 (Experimental): Participants with moderate chronic liver disease enrolled in Part 2 received one 5-mg preladenant tablet, orally, on Day 1.
  Interventions: Drug: Preladenant
- Healthy to Match Moderate HI Part 2 (Active Comparator): Healthy volunteers with normal hepatic function matched to participants with moderate chronic liver disease by race, age, BMI, and gender, enrolled in Part 2 received one 5-mg preladenant tablet, orally, on Day 1.
  Interventions: Drug: Preladenant

INTERVENTIONS:
Drug: Preladenant — After at least an 8 hours overnight fast, one 5-mg preladenant tablet, is administered orally, on Day 1.
  Other Names: SCH 420814; MK-3814; Adenosine 2a Antagonist

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (PK) of preladenant after administration of a single 5 mg oral dose of preladenant in participants with hepatic impairment and healthy volunteers. Part 1 of this study compares healthy volunteers with participants with mild hepatic impairment. Part 2 compares healthy volunteers with participants with moderate hepatic impairment. Healthy volunteers in each part of this study are to be matched with participants with hepatic impairment by race, age, gender, and body mass index (BMI). The primary hypotheses are that in participants with mild or moderate HI, the area under the concentration-time curve from time 0 extrapolated to time of the last quantifiable concentration (AUC0-t) of preladenant is similar to that observed in matched healthy volunteers, so that the mean ratio of hepatic impaired/healthy is contained within the interval [0.50, 2.00].

ELIGIBILITY:
Key Inclusion Criteria for Healthy Participants Groups:

* Must be healthy with normal hepatic function and be free of any clinically significant disease or condition that requires a physician's care and/or would interfere with study evaluations or procedures.

Key Inclusion Criteria for Hepatic Impaired Groups:

* Must have mild or moderate hepatic impairment.
* Must have a diagnosis of chronic liver disease for >6 months.
* Clinical laboratory tests, physical examination, and electrocardiographs must be clinically acceptable to the investigator and sponsor.
* Must be free, other than chronic liver disease, of significant medical conditions unrelated to their hepatic disorder except for conditions that in the opinion of the investigator may not interfere with the study evaluations, procedures or participation.

Key Exclusion Criteria

* Must not be on any prohibited medications for entry into the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-11-10 (Actual); Primary Completion 2012-06-14 (Actual); Study Completion 2012-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate HI Part 2: Participants with moderate chronic liver disease enrolled in Part 2 one 5-mg preladenant tablet, orally, on Day 1.
Period: Overall Study
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Started | 12 | 12 | 9 | 9
Completed | 12 | 12 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2 | Total
Number analyzed (Participants) | 12 | 12 | 9 | 9 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (6.5) | 52.3 (7.1) | 52.2 (4.8) | 50.1 (3.3) | 52.7 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 4 | 4 | 8
  Male | 12 | 12 | 5 | 5 | 34

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Time of the Last Quantifiable Concentration (AUC 0-t) of Preladenant After a Single Dose of Preladenant
Description: For healthy and HI participants blood samples were collected at pre-dose (0 hour) and at 0.50, 1, 2, 4, 6, 12, 16, 24, 30, 36, and 48 hours postdose. Blood samples were also collected for HI participants only at 60 and 72 hours postdose in order to determine the AUC 0-t of preladenant.
Time Frame: Pre-dose up to 72 hours postdose
Population: All participants who received an oral dose of preladenant and for whom at least one pharmacokinetic parameter can be calculated for the treatment phase according to the protocol and who did not have any protocol deviation interfering with pharmacokinetics.
Measure: Least Squares Mean (Full Range); unit: hr*ng/mL
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Number analyzed (Participants) | 12 | 12 | 9 | 9
hr*ng/mL | 97.864 [33.181 to 304.594] | 91.014 [27.457 to 171.810] | 300.667 [81.081 to 571.197] | 115.715 [16.816 to 352.507]
Statistical Analysis 1: Comparison: Mild Hepatic Impaired (HI) Part 1 vs Healthy to Match Mild HI Part 1; The analysis was performed using an analysis of covariance (ANCOVA) model. Parameters were log-transformed (using the natural logarithm) prior to analysis. Study population (i.e., HI or Healthy) was included as a fixed effect with continuous covariates age, Body Mass Index (BMI) and a categorical covariate, gender. Gender was excluded from Part 1 analysis; Test type: Non-Inferiority or Equivalence — To be considered equivalent the least squares mean (LSM) Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.075, 90% CI 2-sided [0.695 to 1.662]
Statistical Analysis 2: Comparison: Moderate HI Part 2 vs Healthy to Match Moderate HI Part 2; The analysis was performed using an ANCOVA model. Parameters were log-transformed (using the natural logarithm) prior to analysis. Study population (i.e., HI or Healthy) was included as a fixed effect with continuous covariates age, BMI and a categorical covariate, gender. Gender was included from Part 2 analysis; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 2.598, 90% CI 2-sided [1.334 to 5.060]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Preladenant After a Single Dose of Preladenant
Description: For healthy and HI participants blood samples were collected at pre-dose (0 hour) and at 0.50, 1, 2, 4, 6, 12, 16, 24, 30, 36, and 48 hours postdose. Blood samples were also collected for HI participants only at 60 and 72 hours postdose in order to determine the Cmax of preladenant.
Time Frame: Pre-dose up to 72 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Full Range); unit: ng/mL
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Number analyzed (Participants) | 12 | 12 | 9 | 9
ng/mL | 39.380 [15.900 to 61.500] | 30.171 [5.890 to 73.200] | 56.997 [8.950 to 109.00] | 39.735 [4.130 to 113.00]
Statistical Analysis 1: Comparison: Mild Hepatic Impaired (HI) Part 1 vs Healthy to Match Mild HI Part 1; The analysis was performed using an ANCOVA model. Parameters were log-transformed (using the natural logarithm) prior to analysis. Study population (i.e., HI or Healthy) was included as a fixed effect with continuous covariates age, BMI and a categorical covariate, gender. Gender was excluded from Part 1 analysis; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.305, 90% CI 2-sided [0.840 to 2.027]
Statistical Analysis 2: Comparison: Moderate HI Part 2 vs Healthy to Match Moderate HI Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.434, 90% CI 2-sided [0.643 to 3.198]

3. Secondary Outcome: AUC 0-t of Preladenant Metabolite SCH 434748 After a Single Dose of Preladenant
Description: For healthy and HI participants blood samples were collected at pre-dose (0 hour) and at 0.50, 1, 2, 4, 6, 12, 16, 24, 30, 36, and 48 hours postdose. Blood samples were also collected for HI participants only at 60 and 72 hours postdose in order to determine the AUC 0-t of SCH 434748.
Time Frame: Pre-dose up to 72 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Full Range); unit: hr*ng/mL
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Number analyzed (Participants) | 12 | 12 | 9 | 9
hr*ng/mL | 28.505 [17.858 to 60.434] | 15.395 [0.156 to 45.462] | 60.486 [17.213 to 96.253] | 25.288 [6.399 to 149.982]
Statistical Analysis 1: Comparison: Mild Hepatic Impaired (HI) Part 1 vs Healthy to Match Mild HI Part 1; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.852, 90% CI 2-sided [0.810 to 4.234]
Statistical Analysis 2: Comparison: Moderate HI Part 2 vs Healthy to Match Moderate HI Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 2.392, 90% CI 2-sided [1.306 to 4.382]

4. Secondary Outcome: Cmax of Preladenant Metabolite SCH 434748 After a Single Dose of Preladenant
Description: For healthy and HI participants blood samples were collected at pre-dose (0 hour) and at 0.50, 1, 2, 4, 6, 12, 16, 24, 30, 36, and 48 hours postdose. Blood samples were also collected for HI participants only at 60 and 72 hours postdose in order to determine the Cmax of SCH 434748.
Time Frame: Pre-dose up to 72 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Full Range); unit: ng/mL
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Number analyzed (Participants) | 12 | 12 | 9 | 9
ng/mL | 10.503 [5.280 to 20.400] | 6.784 [0.624 to 21.400] | 13.983 [4.530 to 52.700] | 9.936 [2.970 to 54.500]
Statistical Analysis 1: Comparison: Mild Hepatic Impaired (HI) Part 1 vs Healthy to Match Mild HI Part 1; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.548, 90% CI 2-sided [0.918 to 2.610]
Statistical Analysis 2: Comparison: Moderate HI Part 2 vs Healthy to Match Moderate HI Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.407, 90% CI 2-sided [0.720 to 2.750]

5. Secondary Outcome: AUC 0-t of Preladenant Metabolite SCH 446637 After a Single Dose of Preladenant
Description: For healthy and HI participants blood samples were collected at pre-dose (0 hour) and at 0.50, 1, 2, 4, 6, 12, 16, 24, 30, 36, and 48 hours postdose. Blood samples were also collected for HI participants only at 60 and 72 hours postdose in order to determine the AUC 0-t of SCH 446637.
Time Frame: Pre-dose up to 72 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Full Range); unit: hr*ng/mL
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Number analyzed (Participants) | 12 | 12 | 9 | 9
hr*ng/mL | 38.262 [18.636 to 87.772] | 24.612 [0.149 to 84.837] | 170.215 [55.366 to 491.013] | 35.421 [10.783 to 70.257]
Statistical Analysis 1: Comparison: Mild Hepatic Impaired (HI) Part 1 vs Healthy to Match Mild HI Part 1; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.555, 90% CI 2-sided [0.617 to 3.917]
Statistical Analysis 2: Comparison: Moderate HI Part 2 vs Healthy to Match Moderate HI Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 4.806, 90% CI 2-sided [2.770 to 8.335]

6. Secondary Outcome: Cmax of Preladenant Metabolite SCH 446637 After a Single Dose of Preladenant
Description: For healthy and HI participants blood samples were collected at pre-dose (0 hour) and at 0.50, 1, 2, 4, 6, 12, 16, 24, 30, 36, and 48 hours postdose. Blood samples were also collected for HI participants only at 60 and 72 hours postdose in order to determine the Cmax of SCH 446637.
Time Frame: Pre-dose up to 72 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Full Range); unit: ng/mL
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Number analyzed (Participants) | 12 | 12 | 9 | 9
ng/mL | 12.691 [6.470 to 29.100] | 10.004 [0.595 to 24.000] | 21.761 [9.840 to 45.600] | 10.993 [4.910 to 21.400]
Statistical Analysis 1: Comparison: Mild Hepatic Impaired (HI) Part 1 vs Healthy to Match Mild HI Part 1; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.269, 90% CI 2-sided [0.703 to 2.288]
Statistical Analysis 2: Comparison: Moderate HI Part 2 vs Healthy to Match Moderate HI Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.980, 90% CI 2-sided [1.316 to 2.977]

7. Secondary Outcome: AUC 0-t of Preladenant Calculated Using Free Drug Concentration After a Single Dose of Preladenant
Description: For healthy and HI participants blood samples were collected at pre-dose (0 hour) and at 0.50, 1, 2, 4, 6, 12, 16, 24, 30, 36, and 48 hours postdose. Blood samples were also collected for HI participants only at 60 and 72 hours postdose in order to determine the AUC 0-t of preladenant calculated using free drug concentration.
Time Frame: Pre-dose up to 72 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Full Range); unit: hr*ng/mL
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Number analyzed (Participants) | 12 | 12 | 9 | 9
hr*ng/mL | 1.605 [0.547 to 6.396] | 1.211 [0.261 to 3.295] | 6.792 [1.133 to 15.708] | 1.681 [0.202 to 6.757]
Statistical Analysis 1: Comparison: Mild Hepatic Impaired (HI) Part 1 vs Healthy to Match Mild HI Part 1; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.326, 90% CI 2-sided [0.749 to 2.348]
Statistical Analysis 2: Comparison: Moderate HI Part 2 vs Healthy to Match Moderate HI Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 4.041, 90% CI 2-sided [1.460 to 11.187]

8. Secondary Outcome: Cmax of Preladenant Calculated Using Free Drug Concentration After a Single Dose of Preladenant
Description: For healthy and HI participants blood samples were collected at pre-dose (0 hour) and at 0.50, 1, 2, 4, 6, 12, 16, 24, 30, 36, and 48 hours postdose. Blood samples were also collected for HI participants only at 60 and 72 hours postdose in order to determine the Cmax of preladenant calculated using free drug concentration.
Time Frame: Pre-dose up to 72 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Full Range); unit: ng/mL
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Number analyzed (Participants) | 12 | 12 | 9 | 9
ng/mL | 0.646 [0.223 to 1.412] | 0.401 [0.130 to 1.129] | 1.288 [0.255 to 2.787] | 0.577 [0.050 to 2.184]
Statistical Analysis 1: Comparison: Mild Hepatic Impaired (HI) Part 1 vs Healthy to Match Mild HI Part 1; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 1.609, 90% CI 2-sided [1.007 to 2.572]
Statistical Analysis 2: Comparison: Moderate HI Part 2 vs Healthy to Match Moderate HI Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — To be considered equivalent the LSM Ratio (HI/Healthy) is contained within the interval [0.50, 2.00]; LSM Ratio = 2.231, 90% CI 2-sided [0.844 to 5.896]

ADVERSE EVENTS:
Time Frame: Up to 7 days
Description: All participants who received an oral dose of preladenant.
Arm/Group | Mild Hepatic Impaired (HI) Part 1 | Healthy to Match Mild HI Part 1 | Moderate HI Part 2 | Healthy to Match Moderate HI Part 2
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 2/12 | 0/12 | 1/9 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hepatic Impaired (HI) Part 1 (N=12) | Healthy to Match Mild HI Part 1 (N=12) | Moderate HI Part 2 (N=9) | Healthy to Match Moderate HI Part 2 (N=9)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with regard to proprietary information; the accuracy of the information; and to ensure that the presentation is fairly balanced and in compliance with Food and Drug Administration (FDA) regulations.